CLINICAL TRIAL: NCT03814018
Title: A Retrospective Study to Verify FEV1 Reversibility Criteria Proposed by the GINA Guidelines, in Asthmatic Children
Brief Title: Bronchoreversibility Test in Asthmatic Children and Correlation With Diagnostic Criteria Proposed by the GINA Guidelines
Acronym: VERI-VEMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0007
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-01

CONDITIONS: Pediatric Asthma
Keywords: Bronchodilation test; GINA; Reversibility criteria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since 2015, GINA (Global INitiative on Asthma) guidelines were modified and adapted to better fit the pediatric population. Asthma diagnosis is mainly based on the results of PFT (Pulmonary Function Tests) and broncho-reversibility test in adult. GINA guidelines modified the requirements to reach a diagnosis of Asthma in children, based on the reversibility test. GINA guideline propose an increase of 12% of the FEV1 is considered as the diagnostic criterium for asthma in pediatrics.

Nevertheless, in clinical practice, most physicians base their diagnosis of asthma in children on the clinical signs presented by the patient and on the efficacy of the prescribed therapy. Also, the spirometric criterium is not sufficiently corroborated by clinical studies. No research has ever looked for the results of bronchoreversibility test in patients receiving a clinical diagnosis of asthma. For this reason, in children with a clinical diagnosis of asthma, the investigators want to look for the results of the bronchoreversibility test and validate that an increase of 12% of the FEV1 correlate with a physician-driven diagnosis of asthma in pediatrics. For further analysis the investigatorswill evaluate also the reversibility of small airways (FEF25-75) and the z-score of the results of the PFT in these children.

ELIGIBILITY:
Inclusion criteria:

* Children aged between 5 and 18 years
* Children with a diagnosis of asthma undergoing a PFT and a bronchoreversibility test on the day of the diagnosis
* Children evaluated at the University Hospital of Montpellier (France), or at the Pediatric Allergy Unit of the University Hospital of Pavia (Italy)

Exclusion criteria:

* Children not able to perform a PFT
* Children taking drugs that could affect the results of a PFT
* Children included in other trials that don't allow them to be included in the present one

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with a physician-base diagnosis of asthma, undergoing a bronchodilation test
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
value of FEV1 increase | 1 day
  Positive predictive value of FEV1 increase (%) in asthmatic children after bronchodilation test
value of FEF 25-75 | 1 day
  Positive predictive value of FEF 25-75 increase (%) in asthmatic children after bronchodilation test

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided